CLINICAL TRIAL: NCT00246441
Title: Paroxetine for Comorbid Social Anxiety Disorder and Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAARAN013379; R01AA013379 (NIH)
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Social Anxiety Disorder; Social Phobia; Alcohol Use Disorder; Alcohol Abuse; Alcohol Dependence
Keywords: Pharmacotherapy; Self medication
MeSH Terms: conditions — Phobia, Social; Alcoholism | interventions — Paroxetine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paroxetine (Experimental): Active medication containing the drug Paroxetine
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator): A Placebo medication that appears just like the active medication but does not contain placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine — 16 weeks treatment; dosing will start at 20 mg/day paroxetine and will increase gradually to a maximum dose of 60 mg/day
  Other Names: paxil
  Arms: Paroxetine
Drug: Placebo — treatment phase will last 16 weeks; dosing will start at 20 mg/day (placebo) and will increase gradually to a maximum dose of 60 mg/day.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether an SSRI, paroxetine, improves social anxiety symptoms and alcohol use in individuals who drink to cope with social anxiety disorder.

DETAILED DESCRIPTION:
Social anxiety disorder (also known as social phobia) is an Axis I anxiety disorder characterized by intense fear and avoidance of social or performance situations in which one might be scrutinized. Its onset is typically in the early teen years. It is the third most common mental disorder in the United States, exceeded in prevalence only by depression and alcoholism. Approximately 20% of the individuals with social anxiety disorder have alcohol problems. Anecdotal and empirical evidence suggests that alcohol is used by some socially anxious individuals to self-medicate anxiety symptoms, a practice that could lead to alcohol abuse and/or dependence. The proposed project further explores the self-medication hypothesis through the use of a double-blind, randomized, placebo-controlled clinical trial. Paroxetine (a selective serotonin reuptake inhibitor) is the drug to be used in the study. Individuals who drink alcohol to cope with social anxiety symptoms and who meet DSM-IV criteria for the dual-diagnoses of social anxiety disorder and alcohol use disorders will be enrolled in the trial. All individuals will be seeking treatment for social anxiety disorder. The treatment phase will last 16 weeks. Dosing will start at 20 mg/day (paroxetine or placebo) and will increase gradually to a maximum dose of 60 mg/day. Each week during treatment and at the end of the trial, assessments will be made with standard instruments to determine the effect of paroxetine (versus placebo) on social anxiety severity, alcohol use, and more specifically, the intentional use of alcohol to cope with social anxiety symptoms. Additionally, 6 month and 12 month follow-up interviews will be conducted. The overarching hypothesis is that because paroxetine will improve social anxiety severity, alcohol use and/or alcohol use for coping will also be reduced in the paroxetine-treated group.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current social anxiety disorder
* Reports social anxiety in most situations (generalized type).
* Treatment seeking for relief of social anxiety.
* Meets DSM-IV criteria for current alcohol use disorder
* Reads at the 6th grade level or above
* Endorses using alcohol to cope with social anxiety either "very often" or "always."
* Reports no prior medical alcohol detoxification
* Willingness to be randomized to the placebo group
* Willingness to attend 16 weekly medication management visits and one alcohol-related therapy session
* Liebowitz Social Anxiety Scale Total score (modified version) of at least 60
* Endorses drinking at least 15 standard drinks in a typical 30 day period or reports drinking heavily (defined as greater-than-or-equal-to 4 standard drinks on one occasion for women; greater-than-or-equal-to 5 standard drinks on one occasion for men, respectively) on at least 2 days in a typical 30 day period.

Exclusion Criteria:

* Abuse or dependence on drugs other than nicotine or marijuana in last 90 days
* Current or past diagnosis of bipolar disorder or schizophrenia
* Significant suicide risk as assessed by the SCID
* Current use of psychotropic medications
* Treatment seeking for alcohol problems
* Any unstable medical condition that might interfere with safe participation in the trial
* Elevated liver enzymes (3 x greater than normal levels)
* History of adverse reaction to paroxetine
* History of failure to respond to adequate trial or dose of paroxetine for social phobia (60 mg/day for at least 6 weeks)
* History of heart problems or abnormal ECG recording
* Pregnancy, nursing, or refusal to use effective birth control if sexually active and premenopausal
* History of one or more alcohol detoxifications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie L Randall, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Paroxetine: Paroxetine
  Paroxetine: 16 weeks treatment; dosing will start at 20 mg/day paroxetine and will increase gradually to a maximum dose of 60 mg/day
- Placebo: Placebo
  Placebo: treatment phase will last 16 weeks; dosing will start at 20 mg/day (placebo) and will increase gradually to a maximum dose of 60 mg/day.
Period: Overall Study
Arm/Group | Paroxetine | Placebo
Started | 20 | 22
Completed | 19 | 22
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine | Placebo | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6.5) | 30 (8.3) | 29 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Social Anxiety Severity
Description: Liebowitz Social Anxiety Scale (LSAS) - each of the two subscales, Fear and Avoidance, each have a maximum possible score of 72 (range 0 to 72). The total score ranges from 0 to 144. A higher score indicates higher severity of Social Anxiety Disorder.
Time Frame: 16 weeks treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine | Placebo
Number analyzed (Participants) | 20 | 22
units on a scale | 87 (14.9) | 93 (18.5)

2. Primary Outcome: Alcohol Use, Quantity and Frequency
Description: Timeline Followback (TLFB), a validated calendar based instrument to assess number of standard drinks consumed on each day of the trial. Baseline measures were computed using past 30 days. From the TLFB, three measures were computed: 1. Proportion of days abstinent (PDA) (the number of days when no drinking occurred, divided by the number of days in the assessment period) (minimum is 0, maximum is 1) (higher score is better), 2. Drinks per drinking day (DDD) (the mean number of standard drinks consumed on a drinking day in the assessment period) (minimum is >0, maximum is infinity) (higher score is worse), 3. Proportion of Heavy Drinking Days (PHD) (the proportion of days each assessment period that a woman consumed 4 or more standard drinks/ man consumed 5 or more standard drinks) (minimum is 0, maximum is 1) (higher score is worse).
Time Frame: 16 weeks treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Paroxetine | Placebo
Number analyzed (Participants) | 20 | 22
units on a scale
  PDA | .66 (.07) | .65 (.07)
  DDD | 5.88 (1.02) | 7.00 (1.48)
  PHD | .54 (.11) | .55 (.13)

3. Primary Outcome: Drinking to Cope
Description: Drinking days that were related to coping with Social Anxiety determined by the TLFB- the proportion of drinking days that were reported to be due to coping with social anxiety. Minimum value is 0, maximum value is 1 Higher is worse.
Time Frame: 16 weeks treatment
Measure: Mean (Standard Error); unit: proportion of drinking days
Arm/Group | Paroxetine | Placebo
Number analyzed (Participants) | 20 | 22
proportion of drinking days | .35 (.1) | .21 (.04)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: We used a 32 item side effect checklist and we asked subjects about all items on the list at each study visit.
Arm/Group | Paroxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 14/20 | 8/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paroxetine (N=20) | Placebo (N=22)
anorgasmia (Reproductive system and breast disorders) | 11 | 4
myoclonus (Musculoskeletal and connective tissue disorders) | 7 | 1
tremor (Nervous system disorders) | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No